CLINICAL TRIAL: NCT05666440
Title: Visco-Circumferential-Suture-Trabeculotomy Versus Rigid Probe Viscotrabeculotomy in Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Assisstant professor of ophthalmology, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCSTvVTinPOAG
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Double armed International study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visco-Circumferential-Suture-Trabeculotomy (Active Comparator): Visco-Circumferential-Suture-Trabeculotomy in Primary Open Angle Glaucoma.
  Interventions: Procedure: Visco-Circumferential-Suture-Trabeculotomy in Primary Open Angle Glaucoma.
- Rigid probe Viscotrabeculotomy (Active Comparator): Rigid probe Viscotrabeculotomy in Primary Open Angle Glaucoma.
  Interventions: Procedure: Rigid probe Viscotrabeculotomy in Primary Open Angle Glaucoma.

INTERVENTIONS:
Procedure: Visco-Circumferential-Suture-Trabeculotomy in Primary Open Angle Glaucoma. — A superior limbal-based conjunctival flap and a paracentesis. A superficial rectangular scleral flap 4×4 mm was fashioned and dissected forward toward the limbus. A deep sceral flap (2×2 mm) was then created toward the limbus underneath the superficial flap exposing the scleral spur and deroofing SC. Viscoelastic (Healon GV, Pfizer, NY) was injected (using a standard 30 G viscocanalostomy cannula) into the ostia of SC Then, the 5/0 polypropylene suture tip was cauterized into a blunt tip (to ensure atraumatic probing of SC). The tip was inserted into the left ostium of SC using a microsurgical forceps and advanced through the whole circumference of the canal. When the tip presented to the right ostium the AC was filled with a viscoelastic through the paracentesis and traction was applied to approximate both ends of the 5/0 polypropylene suture, thus creating a visco-360-degree trabeculotomy.
  Arms: Visco-Circumferential-Suture-Trabeculotomy
Procedure: Rigid probe Viscotrabeculotomy in Primary Open Angle Glaucoma. — A fornixbased conjunctival incision followed by creation of a partial thickness (about 50% thickness) triangular (4×4×4 mm) scleral fap, followed by localization of Schlemm's canal by radial incisions straddling the limbus. High viscosity sodium hyaluronate (Healon GV, Pfzer) was then slowly injected into both ends of Schlemm's canal. Trabeculotomy was completed using the standard Harm's trabeculotome (Geuder Instruments), the scleral fap was then secured tightly with interrupted 10/0 Nylon sutures and conjunctival closure ensued.
  Arms: Rigid probe Viscotrabeculotomy

SUMMARY:
Visco-Circumferential-Suture-Trabeculotomy versus Rigid probe Viscotrabeculotomy in Primary Open Angle Glaucoma.

DETAILED DESCRIPTION:
Introduction Glaucoma is the leading cause of irreversible visual loss worldwide. Primary open angle glaucoma (POAG) is the most common type of glaucoma accounting for 74% of all glaucoma cases (1, 2). Trabeculectomy is still the most commonly performed glaucoma surgery worldwide (3). However, trabeculectomy has several vision-threatening complications as ocular hypotony, choroidal detachment and bleb related infections (4). Therefore, in the recent years, bleb independent less invasive procedures as canaloplasty (5,6), gonioscopy-assisted transluminal trabeculotomy (GATT) (7,8) and ab externo circumferential trabeculotomy (6,9) have become increasingly popular because of their great efficacy and excellent safety profile. Despite the successful outcomes and the few postoperative complications of GATT in juvenile and adult POAG, however on the downside, surgeons with less experience performing GATT procedure may initially struggle with it. Also, GATT requires a goniolens and a reasonably clear cornea to visualize the nasal angle. Introducing instruments into the anterior chamber also poses an increased risk for damage to intraocular structures (10, 11). Looking at ab externo trabeculotomy, for many years, many authors have demonstrated its efficacy in lowering IOP in congenital (12, 13, 14), juvenile (15, 16) and adult open angle glaucomas (6, 9, 17). Trabeculotomy ab externo techniques include conventional probe trabeculotomy, viscotrabeculotomy (VT) (17), 360 - degree suture trabeculotomy (9) , viscocircumferential -suture trabeculotomy (VCST) (14) and trabeculotomy with the use of illuminated microcatheter.(15,18). Although the illuminated microcatheter helps to cannulate SC safely, however its cost constitutes a financial burden in many countries. VCST was proved to be effective for reduction of IOP in PCG as it offers the advantages of performing 360 circumferential trabeculotomy with a great ease and a low cost (14). The aim of the present study was to compare the surgical outcomes of (VCST) and rigid probe VT in patients with POAG.

Purpose:

This study aims to compare the surgical outcomes of (VCST) and rigid probe VT in patients with POAG.

Methods:

The study is conducted at Mansoura university ophthalmic Center. Sample size has been calculated using Cochran's formula with a 95% confidence level and Z value of 1.95. This comparative study was conducted on 166 eyes of 107 patients with medically uncontrolled primary open-angle glaucoma diagnosed and operated upon in the Mansoura Ophthalmic Center of Mansoura University, Egypt between February 2017 and December 2020. The study follows the tenets of the Declaration of Helsinki. All patients of the study received a clear explanation of the study design, the surgical procedures and their possible consequences and they gave written informed consent.

Preoperative Evaluation All of the patients underwent a full ophthalmological examination, particularly estimation of the best corrected visual acuity (BCVA) (the decimal notation was converted to LogMAR), slit lamp examination, IOP measurement by Goldmann's applanation tonometry, gonioscopy using Goldmann 3-mirrors goniolens for angle grading using Schaffer's grading system and fundus examination. Visual field (VF) assessment was performed by SITA strategy perimetry (Humphrey, central 24-2 standard strategy). Retinal nerve fiber layer (RNFL) thickness and optic disc were evaluated using a spectral domain optical coherence tomography (OCT; Topcon, Japan). The number of antiglaucoma medications was recorded.

Eyes with primary open-angle glaucoma, with a gonioscopically open angle, an IOP above 21 mm Hg despite the maximally tolerated antiglaucoma medications, glaucomatous visual field defects, and glaucomatous optic disc appearance, in the absence of any obvious cause for glaucoma, were included in the study.

Patients with primary angle-closure glaucoma, secondary glaucomas, and who were on anticoagulant therapy and cannot stop treatment or with media opacity that interfere with visual field testing or OCT imaging were excluded from the study.

In patients suffering bilateral POAG (59 patients), randomization to either VCST or VT was applied to the first operated eye while the other eye was automatically assigned to the other procedure and included in the study. All surgical procedures were performed by the same experienced surgeon (A.S.E.).

Surgical Technique:

Surgical techniques of both Visco-Circumferential-Suture-Trabeculotomy (VCST) and rigid probe Viscotrabeculotomy (VT) were described previously in details.(14, 17) In Visco-Circumferential-Suture-Trabeculotomy (VCST), exposure of the operative field through a corneal traction suture (vicryl 6/0) placed superiorly was followed by a superior limbal-based conjunctival flap and a paracentesis. After adequate hemostasis, a superficial rectangular scleral flap 4×4 mm was fashioned and dissected forward toward the limbus. A deep sceral flap (2×2 mm) was then created toward the limbus underneath the superficial flap exposing the scleral spur and deroofing SC. Viscoelastic (Healon GV, Pfizer, NY) was gradually injected (using a standard 30 G viscocanalostomy cannula) into the ostia of SC (dilate SC and facilitate suture progression into the canal). Then, the 5/0 polypropylene suture tip was cauterized into a blunt tip (to ensure atraumatic probing of SC). The tip was inserted into the left ostium of SC using a microsurgical forceps and advanced through the whole circumference of the canal. When the tip presented to the right ostium the AC was filled with a viscoelastic through the paracentesis and traction was applied to approximate both ends of the 5/0 polypropylene suture, thus creating a visco-360-degree trabeculotomy.

For the viscotrabeculotomy group, the surgical procedure involved a fornixbased conjunctival incision followed by creation of a partial thickness (about 50% thickness) triangular (4×4×4 mm) scleral fap, followed by localization of Schlemm's canal by radial incisions straddling the limbus. High viscosity sodium hyaluronate (Healon GV, Pfzer) was then slowly injected into both ends of Schlemm's canal. Trabeculotomy was completed using the standard Harm's trabeculotome (Geuder Instruments), the scleral fap was then secured tightly with interrupted 10/0 Nylon sutures and conjunctival closure ensued. For the trabeculectomy group the fornix-based conjunctival incision was followed by mitomycin C application in a concentration of 0.3 mg/mL for 3 min through soaked surgical sponge inserted underneath the conjunctival fap and over the sclera posterior to the limbus then thoroughly irrigated by 200 mL of sterile normal saline. This was followed by dissection of the scleral fap which was rectangular (4×3 mm), followed by trabeculectomy, peripheral iridectomy and then secure closure by 10/0 nylon sutures. Filtration was judged arbitrarily according to the surgeon's experience and the conjunctiva was then closed securely .

For both groups postoperative treatment consisted of topical steroids (dexamethasone) and antibiotic (ofoxacin) five times daily with gradual taper over a 5 week period.

Cycloplegia (cyclopentolate) was used 3 times daily for the first postoperative week and then discontinued. Patients were examined on the first postoperative day and then postoperative follow up visits were scheduled at weeks 1 and 2 then months 1, 2 and 3 and then 3 monthly till the end of the 24th month (months 6, 9, 12, 15, 18, 21 and 24). Complications were noted and managed accordingly. The primary outcome measure was the IOP. Secondary outcome measures included the BCVA and number of IOP lowering medications. Success was defned as [15] an IOP ≤ 18 mmHg (criteria 1), an IOP ≤ 16 mmHg (criteria 2), IOP ≤ 14 mmHg (criteria 3) and ≤ 12 mmHg (criteria 4) and/or IOP reduction by ≥ 30% of baseline IOP (last IOP measurement immediately before surgery) without IOP lowering medications (complete success) (qualifed success was defned as IOP controlled according to the same criteria with/without IOP lowering medications), without the need for further surgery for IOP reduction and without any vision threatening complications or hypotony (IOP ≤ 5 mmHg).

Statistical analysis:

Data were analysed with IBM SPSS. Repeated measure ANOVA and paired t tests were used to compare the preoperative and postoperative variables in each group. Assessment of the data normality will be done using both histogram plot and Shapiro-Wilk's test. The comparison between the two groups was done by Independent samples T test for numerical variables and Chi-square test for categorical variables. Fisher's exact p values were chosen where there was an expected count of less than 5. Kaplan-Meier survival curves were plotted to estimate the mean survival time and probabilities of failure at diferent follow-up stages in the both groups.. For all tests, P value of less than 0.05 will be considered significant.

References

1. Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol 2006;90:262 7. 10.1136/bjo.2005.081224.
2. Kapetanakis VV, Chan MP, Foster PJ, Cook DG, Owen CG, Rudnicka AR. Global variations and time trends in the prevalence of primary open angle glaucoma (POAG): a systematic review and meta-analysis. Br J Ophthalmol. 2016 Jan;100(1):86-93. doi: 10.1136/bjophthalmol-2015-307223. Epub 2015 Aug 18.PMID: 26286821; PMCID: PMC4717368.
3. Jed L, Goldberg I. Current management of glaucoma. Med J Aust. 2019;210:180-187.
4. Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC; Tube Versus Trabeculectomy Study Group. Postoperative complications in the Tube Versus Trabeculectomy (TVT) study during five years of follow-up. Am J Ophthalmol. 2012;153(5):804-14 e1.
5. Riva I, Brusini P, Oddone F, Michelessi M, Weinreb RN, Quaranta L. Canaloplasty in the Treatment of Open-Angle Glaucoma: A Review of Patient Selection and Outcomes. Adv Ther. 2019 Jan;36(1):31-43. doi: 10.1007/s12325-018-0842-6. Epub 2018 Nov 28. PMID: 30488337; PMCID: PMC6318242.
6. Wang H, Xin C, Han Y, Shi Y, Ziaei S, Wang N. Intermediate outcomes of ab externo circumferential trabeculotomy and canaloplasty in POAG patients with prior incisional glaucoma surgery. BMC Ophthalmol. 2020 Oct 2;20(1):389. doi:10.1186/s12886-020-01645-0. PMID: 33008405; PMCID: PMC7531087.
7. Aktas Z, Ucgul AY, Bektas C, Sahin Karamert S. Surgical Outcomes of Prolene Gonioscopy-assisted Transluminal Trabeculotomy in Patients With Moderate to Advanced Open-Angle Glaucoma. J Glaucoma. 2019 Oct;28(10):884-888. doi: 10.1097/IJG.0000000000001331. PMID: 31385914.
8. Faria BM, Daga FB, Rebouças-Santos V, Araújo RB, Matos Neto C, Jacobina JS,Faria MAR. Gonioscopy-assisted transluminal trabeculotomy (GATT) outcomes in eyes with open-angle glaucoma resistant to maximum treatment. Arq Bras Oftalmol. 2021 Nov-Dec;84(6):587-593. doi: 10.5935/0004-2749.20210083. PMID: 34320113.
9. Yalinbas D, Dilekmen N, Hepsen IF. Comparison of Ab Externo and Ab Interno 360-degree Suture Trabeculotomy in Adult Open-angle Glaucoma. J Glaucoma. 2020 Nov;29(11):1088-1094. doi: 10.1097/IJG.0000000000001627. PMID: 32769730.
10. Rahmatnejad K., Pruzan N.L., Amanullah S., Shaukat B.A., Resende A.F.,Waisbourd M., Zhan T., Moster M.R. Surgical Outcomes of Gonioscopy-assisted Transluminal Trabeculotomy (GATT) in Patients with Open-angle Glaucoma. J.Glaucoma. 2017;26:1137-1143. doi: 10.1097/IJG.0000000000000802.
11. Grover D.S., Smith O., Fellman R.L., Godfrey D.G., Gupta A., Montes de Oca I., Feuer W.J. Gonioscopy-assisted Transluminal Trabeculotomy: An Ab Interno Circumferential Trabeculotomy: 24 Months Follow-up. J. Glaucoma.2018;27:393-401. doi: 10.1097/IJG.0000000000000956.
12. Filous A, Brunová B. Results of the modified trabeculotomy in the treatment of primary congenital glaucoma. J AAPOS. 2002 Jun;6(3):182-6. doi:

    10.1067/mpa.2002.123431. PMID: 12075295.
13. Elwehidy AS, Hagras SM, Bayoumi N, AbdelGhafar AE, Badawi AE. Five-year results of viscotrabeculotomy versus conventional trabeculotomy in primary congenital glaucoma: A randomized controlled study. Eur J Ophthalmol. 2021Mar;31(2):786-795. doi: 10.1177/1120672120922453. Epub 2020 May 26.PMID: 32450720.
14. Elwehidy AS, Bayoumi NHL, Abd Elfattah D, Hagras SM. Surgical Outcomesof Visco-Circumferential-Suture-Trabeculotomy Versus Rigid Probe

    Trabeculotomy in Primary Congenital Glaucoma: A 3-Year RandomizedControlled Study. J Glaucoma. 2022 Jan 1;31(1):48-53. doi:

    10.1097/IJG.0000000000001944. PMID: 34628421.
15. Dao JB, Sarkisian SR Jr, Freedman SF. Illuminated microcatheter-facilitated 360-degree trabeculotomy for refractory aphakic and juvenile open-angle glaucoma. J Glaucoma. 2014 Sep;23(7):449-54. doi:10.1097/IJG.0b013e31829484df. PMID: 23661045.
16. Lim ME, Dao JB, Freedman SF. 360-Degree Trabeculotomy for Medically Refractory Glaucoma Following Cataract Surgery and Juvenile Open-Angle Glaucoma. Am J Ophthalmol. 2017 Mar;175:1-7. doi:10.1016/j.ajo.2016.11.011. Epub 2016 Dec 1. PMID: 27916715.
17. Elwehidy AS, Mokbel TH, Bayoumi NHL, Badawi AE, Hagras SM. Viscotrabeculotomy versus trabeculectomy in the surgical treatment of open angle glaucoma: a single center, randomised controlled trial. Jpn J Ophthalmol.2021 May;65(3):395-401. doi: 10.1007/s10384-020-00801-9. Epub 2021 Jan 7.PMID: 33415606.
18. Zhang W, Wang Y, Xin C, Sun Y, Cao K, Wang H, Wang N. Ab Interno vs. Ab Externo Microcatheter-Assisted Circumferential Trabeculotomy in Treating Patients With Primary Open-Angle Glaucoma. Front Med (Lausanne). 2021 Dec 20;8:795172. doi: 10.3389/fmed.2021.795172. PMID: 34988099; PMCID: PMC8720850.

ELIGIBILITY:
Inclusion Criteria:

- The diagnosis of OAG was based on the optic nerve head appearance typical to glaucoma (increased optic disc cupping, thinning of the neuro-retinal rim, focal notching, splinter haemorrhage), corresponding visual feld loss typical to glaucoma coupled with an elevated IOP above the statistical normal of 21 mmHg and a gonioscopically open angle in the absence of any known cause for glaucoma. IOP-lowering medications were initiated for all patients and only those patients in whom control of the disease failed (as evidenced by progressive optic nerve damage and/or visual feld deterioration) and the decision for surgical intervention to lower the IOP was taken were enrolled in the study. Adult patients (above 18 years of age) fulflling these criteria were enrolled

Exclusion Criteria:

Other types of glaucomas and co-morbidities

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure was the IOP | 2 years
  Success was defned as [15] an IOP ≤ 18 mmHg (criteria 1), an IOP ≤ 16 mmHg (criteria 2), IOP ≤ 14 mmHg (criteria 3) and ≤ 12 mmHg (criteria 4) and/or IOP reduction by ≥ 30% of baseline IOP (last IOP measurement immediately before surgery) without IOP lowering medications (complete success) (qualifed success was defned as IOP controlled according to the same criteria with/without IOP lowering medications), without the need for further surgery for IOP reduction and without any vision threatening complications or hypotony (IOP ≤ 5 mmHg).
BCVA | 2 years
number of IOP lowering medications. | 2 years

IPD SHARING:
Plan to Share IPD: Yes
supplemental digital content
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code